CLINICAL TRIAL: NCT01916720
Title: A Multi-centre, Randomised, Double-blind, Placebo-controlled, Parallel-group Study to Investigate the Effect of the Lp-PLA2 Inhibitor SB-480848 (40, 80mg od) on Carotid Plaque Composition in Patients With Carotid Artery Disease and Planned Carotid Endarterectomy, Stratified for Statin Use and Gender, After 14+/-4 Days Treatment
Brief Title: Study to Determine the Effect of 14 Days Dosing With Darapladib (SB-480848) on Carotid Plague Composition in Patients With Planned Carotid Endarterectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 480848/010
Record Dates: First submitted 2013-07-31; First posted 2013-08-06 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — darapladib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- SB-480848 40 mg (Experimental): SB-480848 40 milligrams (mg) once a day (od) for 14 +/- 4 days followed by carotid endarterectomy. SB-480848 40 mg was administered as 2 SB-480848 20 mg tablets plus 2 placebo tablets.
  Interventions: Drug: SB-480848 40 mg; Drug: Placebo
- SB-480848 80 mg (Experimental): SB-480848 80 mg od for 14 +/- 4 days followed by carotid endarterectomy.SB-480848 80 mg was administered as 4 20 mg SB-480848 tablets.
  Interventions: Drug: SB-480848 80 mg
- Matching Placebo (Placebo Comparator): Placebo for 14 +/- 4 days followed by carotid endarterectomy. Placebo was administered as 4 placebo tablets. Placebo tablets were identical in appearance to the SB-480848 20 mg tablets.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SB-480848 40 mg — Study Drug
  Arms: SB-480848 40 mg
Drug: SB-480848 80 mg — Study Drug
  Arms: SB-480848 80 mg
Drug: Placebo — Study Drug
  Arms: Matching Placebo; SB-480848 40 mg

SUMMARY:
The primary objective is to determine Lp-PLA2 activity in atherosclerotic carotid plaques after 14 (+/-4) days treatment with darapladib, compared to placebo. Secondary objectives include determination of the change in Lp-PLA2 activity in blood, Lp-PLA2 mass in blood and plaque, specified biomarkers in blood and plaque and their respective correlation's with Lp-PLA2. In addition, the study aims to characterise the PK/PD of repeat oral doses of SB-480848, and safety and tolerability in this population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, >35 years of age
* Females of childbearing potential must be using approved contraceptive measures
* Male patients must be willing to abstain from sexual intercourse or use a form of contraception if engaging in sexual intercourse with a woman who could become pregnant
* Planned carotid endarterectomy within a timeframe compatible with recruitment for the study and able to comply with the requirements of the study, as deemed by the investigator
* Written, informed consent to participate

Exclusion Criteria:

* Recent myocardial infarction (within the previous 4 weeks)
* Currently taking corticosteroids, warfarin, digoxin or a potent CYP3A4 inhibitor
* Recent (<3 months) or ongoing acute infection or significant trauma associated with bruising and/or taking antibiotics. Prophylactic antibiotics for surgery are allowed
* Change in dose of lipid-lowering therapy during the previous 4 weeks from randomisation
* History of chronic liver disease (e.g. cirrhosis, hepatitis) OR ALT OR AST ≥1.5 times the upper limit of normal (ULN) at screening
* Diagnosis of systemic lupus erythematosis (SLE) or rheumatoid arthritis (RA)
* Clinically significant anaemia
* History of severe renal impairment (serum creatinine >1.8mg/dL)
* Unstable angina
* History of asthma , anaphylaxis or anaphylactoid reactions, severe allergic responses
* Abuse of alcohol or drugs within the last 6 months
* Any factor or clinical disease state that, in the investigator's opinion, would preclude completion of a safe surgical procedure and/or completion of the study
* Use of an investigational drugs within 30 days or 5 half-lives of their last dose prior to starting the study, whichever is the longest

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2003-01; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Lp-PLA2 activity in the atherosclerotic plaque removed during carotid endarterectomy | 14 +/- 4 days

SECONDARY OUTCOMES:
Lp-PLA2 mass in plaque removed during the carotid endarterectomy | 14 +/- 4 days
Lp-PLA2 mass and activity in blood | 14 +/- days
Lipid and Non-Lipid Biomarkers in Plasma | 14 +/- days
  Lipids: total cholesterol, HDL, LDL, and triglycerides Non-Lipids: hsCRP, CD40L, ICAM-1, E-selectin, PAI-1 antibody, PAI-1 antigen, and MMP-9
Oxidised Lipids and Their Metabolites, and Biomarkers in Plaque | 14 +/- 4 days
  Oxidised Lipids and Their Metabolites: total lyso-PC, total phospholipid, and total phosphatidylcholine Biomarkers: CD68 (macrophages), CD3 (T cells), CD20 or CD22 (B cells), alpha-actin (smooth muscle cells), CD40L, MMP-2, MMP-9, PAI-1, ICAM-1, IL-6, and Lp-PLA2 (mRNA expression)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Johnson JL, Shi Y, Snipes R, Janmohamed S, Rolfe TE, Davis B, Postle A, Macphee CH. Effect of darapladib treatment on endarterectomy carotid plaque lipoprotein-associated phospholipase A2 activity: a randomized, controlled trial. PLoS One. 2014 Feb 20;9(2):e89034. doi: 10.1371/journal.pone.0089034. eCollection 2014. PMID 24586490
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 480848/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 480848/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 480848/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 480848/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 480848/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 480848/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 480848/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register